CLINICAL TRIAL: NCT02783326
Title: Effects of a Protocol Of Rehabilitation in Patients With Chronic Disease Obstructive Pulmonary (COPD) Improvement Modulation Autonomic Heart Rate, Oxidative Stress, Quality of Life and Function
Brief Title: Rehabilitation Cardiorrespiratory Improvement in Patients With Chronic Disease Obstructive Pulmonary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Principal investigator, Universidade Metodista de Piracicaba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1322578
Record Dates: First submitted 2016-03-11; First posted 2016-05-26 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Chronic Disease Obstructive Pulmonary
Keywords: Chronic Disease Obstructive Pulmonary; Rehabilitation; Physical Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPD Group (Experimental): Evaluation of oxidative stress, heart rate variability, quality of life with AQ20 questionary, function with TC6 before the application of rehabilitation protocol, after 10 weeks during protocol application and 2 months after protocol application
  Interventions: Other: Rehabilitation
- Control Group (Active Comparator): Evaluation of oxidative stress, heart rate variability, quality of life with AQ20 questionary, function with TC6 before the application of rehabilitation protocol, after 10 weeks during protocol application and 2 months after protocol application
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Pulmonary rehabilitation, exercise in COPD individuals and health individuals

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a condition in which the lung is in chronic state due to an inflammatory response that leads to limitation in lung function of the individual, providing symptoms such as dyspnea, nutritional changes, decreased strength respiratory muscle, low capacity to exercise, dynamic insufflation and altered autonomic function with decreased heart rate variability. Have objective to evaluate and compare the effects of a rehabilitation protocol on autonomic modulation of heart rate. Participate in the study, 10 volunteers with COPD and 10 apparently healthy individuals, of both sexes, between 50 and 70 years old. Data collection and application of the Protocol will take place at the Clinical School of Physiotherapy and Occupational Therapy at the University of the Amazon (UNAMA). Between January and February 2015.

DETAILED DESCRIPTION:
The study is being conducted in the physiotherapy clinic of HUJBB. The sample is composed of 26 volunteers with moderate to severe COPD, of both genders, recruited from the population that will start the treatment in pulmonology HUJBB physiotherapy clinic.

All participants will undergo the assessment base used in HUJBB, blood analysis, heart rate variability, AQ20 questionary, 6-minute walk test and Pulmonary Rehabilitation Program.

The evaluation will be carried out by pre-existing general assessment form and used in hospital outpatient. The sheet contains: identification data; medical history; diagnosed diseases; Drug use; Use of oxygen; nutrition and exercise habits; Physical exam; Investigations; functional kinetic evaluation; Goals; treatment/management. Since these will only be used: identification data; diagnosed diseases; Use of Oxygen; nutrition and exercise habits and goals.

Morphological assessment of EOX in blood plasma is performed according to the test known as Optical Microscopy for cell analysis in vitro or HLB test, also known under the name Dry layer oxidative test, which the investigators refer to as microscopic morphology EOX in plasma (EEW). The EEW provides indirect information concerning EOX, among others, using the following grading system percentage of discontinuous area of the clot, present in the microscope slide: grade I (normal EOX rate, with total area of discontinuity of the extracellular matrix (ME) less than 10%), grade II (light EOX with ME discontinuity area between 10 to 20%), grade III (moderate EOX with ME discontinuity area between 20 to 30%), grade IV ( serious EOX with ME discontinuity area between 30 to 40%) and the grade V (very serious EOX with ME discontinuity area above 40%) 18. By lancing on the medial side of the digital pulp of the fourth finger of the left hand previously sanitized with alcohol, collecting the blood drop will be next to a microscope slide by five light touches this blade with the drop. After this procedure, the blade will be kept in place protected from contact with the blood and at room temperature (23 ° C) for the nine-minute period for the realization of the collected blood clotting process. At the end of this period, the morphological patterns of these clots are seen in an increase of 40 times as set out in protocolo18 and their assigned qualitative graduation will be logged into a spreadsheet for further statistical analysis.

The coagulated blood will be studied by Videomicroscopy (microscope NIPOM brand), which will be selected the best histological field, then a picture which will be analyzed by Image Pro Plus you see the fields where there is no blood coagulation will be made, and from this discontinuity the program will provide the percentage of oxidative stress. This analysis test allows you to have an indirect notion of oxidative stress level in the studied patient and to evaluate its therapeutic development.

The uptake of HRV is performed via a heart rate monitor Polar ® brand of, RS800CX model where the FC signal is received by a strap to the signal receiver which is placed in the voluntary thorax at the level of the xiphoid the sternum. This funding is recorded in the Polar RS800CX monitor and transferred to the Software Polar ProTrainer program through a broadcast interface infrared signals, which are stored and subsequently exported to txt format so that later can be analyzed by a mathematical routine in Kubios HRV program. In the program will be selected 5 minutes from the passage that has better signal stability.

HRV will be analyzed at rest in the supine position. This test is to evaluate the variability of the heart rate response to check the modulation of autonomic control over it at rest in the supine position.

Volunteers will be asked to remain at rest for a period of 10 minutes, avoiding talking to the researcher so that the heart rate does not undergo changes. Then will begin the collection of heart rate with duration of 10 minutes in the supine position while maintaining spontaneous breathing.

The AQ20 is applied twice to the same patient, once in the first day and a second time after the end of the program. Only two researchers participated in the questionnaire.

The hall used to perform the 6MWT should have a comfortable temperature, and can be a closed or outdoor environment, since it is flat, and little traveled so there are no interruptions while walking by people who move there. Usually you use a corridor 30 meters long, with no obstacles where the time to make a turn must be marked with a cone. The test objective is to walk in itself alone pace as far as possible during the six minutes and guiding possible cardiorespiratory changes that may arise, being allowed to walk slowly, stop, relax when needed returning to walk when you feel able to resume the walk. You must walk without talking to the people who are around you to the cone and will back quickly around it so continuing to walk without hesitation. The path must be shown to the patient by the examiner and can start walking.

The training will run 2 times a week (Monday and Wednesday or Tuesday and Thursday ), lasting approximately 50 minutes of specific training ( aerobic and strengthening), for 10 weeks, making a total of 20 days of exercise.

During this period volunteers will be told not to perform complementary physical activities and/or addition to another rehabilitation program.

strengthening exercises involve large muscle groups of the regions of the shoulder, knee and hip in closed and open chain using the Neuromuscular Facilitation ( PNF) with upper extremity exercises within the movements of the diagonals of Kabat method (flexion -adduction -rotation external / foreign flexion - abduction -rotation / internal extension - abduction - rotation / internal extension - adduction - rotation ). The exercises follow the protocol 3 sets of 10 repetitions at intervals of 30 seconds of rest.

ELIGIBILITY:
Inclusion Criteria:

* individuals who have been diagnosed with COPD , stage II and III disease
* are undergoing treatment at the hospital João de Barros Barreto in the period January and February 2016
* both sexes
* 50 to 70 years of age
* hemodynamically stable

Exclusion Criteria:

* were not diagnosed with COPD
* present associated diseases that may interfere with cardiac autonomic control,
* had less than 50 years or over 70 years old
* are in stage I of the COPD
* in intensive care unit
* present muscle skeletal deformities
* hemodynamic instability
* make use of pacemakers
* in need of supplemental O2
* who do not tolerate the practice of exercises

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Heart rate variability modulation | Change from baseline autonomic modulation at 2 months
  Heart rate variability evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo S Rocha, Master, Principal Investigator — Universidade Metodista de Piracicaba
Locations (1):
- Hospital João de Barros Barretos, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Borghi-Silva A, Arena R, Castello V, Simoes RP, Martins LE, Catai AM, Costa D. Aerobic exercise training improves autonomic nervous control in patients with COPD. Respir Med. 2009 Oct;103(10):1503-10. doi: 10.1016/j.rmed.2009.04.015. Epub 2009 May 22. PMID 19464865
- [Result] Fischer BM, Pavlisko E, Voynow JA. Pathogenic triad in COPD: oxidative stress, protease-antiprotease imbalance, and inflammation. Int J Chron Obstruct Pulmon Dis. 2011;6:413-21. doi: 10.2147/COPD.S10770. Epub 2011 Aug 5. PMID 21857781
- [Result] Decramer M. Response of the respiratory muscles to rehabilitation in COPD. J Appl Physiol (1985). 2009 Sep;107(3):971-6. doi: 10.1152/japplphysiol.91459.2008. Epub 2009 Apr 2. PMID 19342436
- [Result] Pelegrino NR, Lucheta PA, Sanchez FF, Faganello MM, Ferrari R, Godoy Id. Influence of lean body mass on cardiopulmonary repercussions during the six-minute walk test in patients with COPD. J Bras Pneumol. 2009 Jan;35(1):20-6. doi: 10.1590/s1806-37132009000100004. English, Portuguese. PMID 19219327
- [Result] Eisner MD, Blanc PD, Sidney S, Yelin EH, Lathon PV, Katz PP, Tolstykh I, Ackerson L, Iribarren C. Body composition and functional limitation in COPD. Respir Res. 2007 Jan 29;8(1):7. doi: 10.1186/1465-9921-8-7. PMID 17261190